CLINICAL TRIAL: NCT01406938
Title: A Randomized, Double-blind, Multicenter Study of Subcutaneous Secukinumab, Assessing Psoriasis Area and Severity Index (PASI) Response and Maintenance of Response in Subjects With Moderate to Severe Chronic Plaque-type Psoriasis on Either a Fixed Dose Regimen or on a Retreatment at Start of Relapse Regimen
Brief Title: Efficacy and Safety of Subcutaneous Secukinumab (AIN457) for Moderate to Severe Chronic Plaque-type Psoriasis Assessing Different Doses and Dose Regimens
Acronym: SCULPTURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457A2304; 2011-000767-27 (EudraCT Number)
Record Dates: First submitted 2011-07-12; First posted 2011-08-01 (Estimated); Results first posted 2015-05-19 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-04

CONDITIONS: Moderate to Severe Plaque-type Psoriasis
Keywords: Psoriasis; plaque; inflammatory skin disease; scaly patches; AIN457; secukinumab; Moderate to Severe Plaque-type Psoriasis
MeSH Terms: conditions — Psoriasis; Plaque, Amyloid; Dermatitis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- AIN457150 mg- Induction period Only(IPO) (Experimental): secukinumab 150 mg (1 injection per dose) and placebo to secukinumab 150 mg (1 injection per dose). Induction period only (IPO)
  Interventions: Drug: AIN457 150mg
- AIN457 300 mg - IPO (Experimental): secukinumab- 2 x 150mg injections per dose
  Interventions: Drug: AIN457 300mg
- AIN457 150 mg - Fixed Interval (FI) (Experimental): 1 s.c. secukinumab 150 mg injection + 1 s.c. PBO (placebo) secukinumab injection
  Interventions: Drug: AIN457 150mg
- AIN457 300 mg FI (Experimental): 2 s.c. secukinumab 150 mg injections
  Interventions: Drug: AIN457 300mg
- AIN457 150 mg- Start of relapse (SoR) (Experimental): 1 s.c. secukinumab 150 mg injection + 1 s.c. PBO secukinumab injection
  Interventions: Drug: AIN457 150mg
- AIN457 300 mg- SoR (Experimental): 2 s.c. secukinumab 150 mg injections
  Interventions: Drug: AIN457 300mg

INTERVENTIONS:
Drug: AIN457 150mg — (1 injection per dose) and placebo to secukinumab 150 mg
  Other Names: secukinumab 150 mg
  Arms: AIN457 150 mg - Fixed Interval (FI); AIN457 150 mg- Start of relapse (SoR); AIN457150 mg- Induction period Only(IPO)
Drug: AIN457 300mg — secukinumab 150 mg (2 injections per dose)
  Other Names: secukinumab
  Arms: AIN457 300 mg - IPO; AIN457 300 mg FI; AIN457 300 mg- SoR

SUMMARY:
This study will assess the safety and efficacy of two different doses and two different dose regimens of subcutaneous secukinumab in patients that have moderate to severe, chronic, plaque-type psoriasis.

ELIGIBILITY:
Inclusion criteria:

* Moderate and severe plaque-type psoriasis diagnosed for at least 6 months.

Severity of disease meeting all of the following three criteria:

* PASI score of 12 or greater,
* Investigator's Global Assessment (IGA) score of 3 or greater
* Total body surface area (BSA) affected of 10% or greater.
* Inadequate control by prior use of topical treatment, phototherapy and/or systemic therapy.

Exclusion criteria:

* Current forms of psoriasis other than chronic plaque-type psoriasis (for example, pustular, erythrodermic, guttate).
* Current drug-induced psoriasis.
* Previous use of secukinumab or any drug that targets IL-17 or IL-17 receptor.
* Significant medical problems such as uncontrolled hypertension, congestive heart failure or a condition that significantly immunocompromises the subject.
* Hematological abnormalities.
* History of an ongoing, chronic or recurrent infectious disease, or evidence of untreated tuberculosis.
* History of lymphoproliferative disease or history of malignancy of any organ system within the past 5 years.
* Pregnant or nursing (lactating) women.
* Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 967 (Actual)
Dates: Start 2011-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (120):
- United States (31):
  - Novartis Investigative Site, Fresno, California
  - Novartis Investigative Site, Pasadena, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Naples, Florida
  - Novartis Investigative Site, South Miami, Florida
  - Novartis Investigative Site, West Palm Beach, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Champaign, Illinois
  - Novartis Investigative Site, Skokie, Illinois
  - Novartis Investigative Site, Springfield, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Overland Park, Kansas
  - Novartis Investigative Site, Owensboro, Kentucky
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Fridley, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Henderson, Nevada
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Verona, New Jersey
  - Novartis Investigative Site, Greensboro, North Carolina
  - Novartis Investigative Site, High Point, North Carolina
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Anderson, South Carolina
  - Novartis Investigative Site, Greer, South Carolina
  - Novartis Investigative Site, Goodlettsville, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
- Austria (4):
  - Novartis Investigative Site, Wels, Austria
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- Bulgaria (4):
  - Novartis Investigative Site, Sofia, Bulgaria
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Canada (5):
  - Novartis Investigative Site, Barrie, Ontario
  - Novartis Investigative Site, Oakville, Ontario
  - Novartis Investigative Site, Waterloo, Ontario
  - Novartis Investigative Site, Windsor, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Czechia (6):
  - Novartis Investigative Site, Brno-Bohunice, Czech Republic
  - Novartis Investigative Site, Hradec Králové, CZE
  - Novartis Investigative Site, Prague, CZE
  - Novartis Investigative Site, České Budějovice
  - Novartis Investigative Site, Nový Jičín
  - Novartis Investigative Site, Prague
- France (5):
  - Novartis Investigative Site, Toulouse, France
  - Novartis Investigative Site, Antony
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Pierre-Benite Cédex
  - Novartis Investigative Site, Rouen
- Germany (20):
  - Novartis Investigative Site, Münster, Germany
  - Novartis Investigative Site, Bad Wildbad
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Buchholz I. D. Nordheide
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dippoldiswalde-Schmiedeberg
  - Novartis Investigative Site, Duisburg
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Mahlow
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Pommelsbrunn
  - Novartis Investigative Site, Wuppertal
- India (7):
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Secunderabad, Andhra Pradesh
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Mangalore, Karnataka
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Nashik, Maharashtra
- Italy (3):
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Verona, VR
- Japan (14):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kisarazu, Chiba
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Asahikawa, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Shimotsuke, Tochigi
  - Novartis Investigative Site, Chiyoda-ku, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
- Poland (3):
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Wroclaw
- Novartis Investigative Site, Singapore, Singapore, Singapore
- Slovakia (6):
  - Novartis Investigative Site, Košice, Slovak Republic
  - Novartis Investigative Site, Košice, Slovakia
  - Novartis Investigative Site, Poprad, Slovakia
  - Novartis Investigative Site, Svidník, Slovakia
  - Novartis Investigative Site, Žilina, Slovakia
  - Novartis Investigative Site, Bratislava
- Switzerland (3):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Zurich
- United Kingdom (5):
  - Novartis Investigative Site, London, England
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Blackpool
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, Poole
- Vietnam (3):
  - Novartis Investigative Site, Hanoi, Vietnam
  - Novartis Investigative Site, Hanoi
  - Novartis Investigative Site, Ho Chi Minh City

REFERENCES:
- [Derived] Merola JF, McInnes IB, Deodhar AA, Dey AK, Adamstein NH, Quebe-Fehling E, Aassi M, Peine M, Mehta NN. Effect of Secukinumab on Traditional Cardiovascular Risk Factors and Inflammatory Biomarkers: Post Hoc Analyses of Pooled Data Across Three Indications. Rheumatol Ther. 2022 Jun;9(3):935-955. doi: 10.1007/s40744-022-00434-z. Epub 2022 Mar 19. PMID 35305260
- [Derived] Dehlin M, Fasth AER, Reinhardt M, Jacobsson LTH. Impact of psoriasis disease activity and other risk factors on serum urate levels in patients with psoriasis and psoriatic arthritis-a post-hoc analysis of pooled data from three phase 3 trials with secukinumab. Rheumatol Adv Pract. 2021 Feb 18;5(1):rkab009. doi: 10.1093/rap/rkab009. eCollection 2021. PMID 33748660

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 966 patients randomized to two groups, induction secukinumab 150 mg or secukinumab 300 mg. Most randomized patients, 928/966 completed the 12-week induction period. 928 completed the induction period, a total of 843 were re-randomized to the maintenance period to either fixed interval dosing or start of relapse dosing at their respective dose level
Period: Induction Period
Arm/Group | AIN457150 mg- Induction Period Only(IPO) | AIN457 300 mg - IPO | AIN457 150 mg - Fixed Interval (FI) | AIN457 300 mg FI | AIN457 150 mg- Start of Relapse (SoR) | AIN457 300 mg- SoR
Started | 482 | 484 | 0 | 0 | 0 | 0
FAS:Patients Assigned Study Treatment | 482 | 483 | 0 | 0 | 0 | 0
Completed | 464 | 464 | 0 | 0 | 0 | 0
Not Completed | 18 | 20 | 0 | 0 | 0 | 0
Not completed — Subject/guardian decision | 6 | 8 | 0 | 0 | 0 | 0
Not completed — Protocol deviation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 8 | 9 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 3 | 0 | 0 | 0 | 0
Period: Maintenance Period
Arm/Group | AIN457150 mg- Induction Period Only(IPO) | AIN457 300 mg - IPO | AIN457 150 mg - Fixed Interval (FI) | AIN457 300 mg FI | AIN457 150 mg- Start of Relapse (SoR) | AIN457 300 mg- SoR
Started | 0 | 0 | 203 | 217 | 206 | 217
FAS: Patients Assigned Treatment Drug | 0 | 0 | 203 | 216 | 206 | 217
Completed | 0 | 0 | 186 | 199 | 181 | 201
Not Completed | 0 | 0 | 17 | 18 | 25 | 16
Not completed — Adverse Event | 0 | 0 | 2 | 8 | 4 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Subject/guardian decision | 0 | 0 | 11 | 7 | 10 | 7
Not completed — Protocol Violation | 0 | 0 | 2 | 2 | 2 | 2
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 4 | 0
Not completed — Lack of Efficacy | 0 | 0 | 2 | 1 | 3 | 5
Period: Follow up
Arm/Group | AIN457150 mg- Induction Period Only(IPO) | AIN457 300 mg - IPO | AIN457 150 mg - Fixed Interval (FI) | AIN457 300 mg FI | AIN457 150 mg- Start of Relapse (SoR) | AIN457 300 mg- SoR
Started | 26 | 23 | 40 | 39 | 40 | 35
Completed | 18 | 18 | 32 | 36 | 31 | 32
Not Completed | 8 | 5 | 8 | 3 | 9 | 3
Not completed — Lack of Efficacy | 3 | 2 | 1 | 0 | 0 | 0
Not completed — Patient/guardian decision | 4 | 2 | 4 | 2 | 4 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 2 | 0 | 3 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The Full analysis set (FAS) was comprised of all patients to whom study treatment had been assigned.
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457150 mg- Induction Period Only(IPO) | AIN457 300 mg - IPO | Total
Number analyzed (Participants) | 482 | 484 | 966
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.3 (12.83) | 46.7 (12.83) | 46.0 (12.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 177 | 151 | 328
  Male | 305 | 333 | 638

OUTCOME MEASURES:

1. Primary Outcome: For the Fixed Interval Group and the Start of Relapse (SoR) Group, the Percentage of Participants (Who Responded to Treatment at Week 12) Maintaining a 75% Improvement From Baseline in Psoriasis Area and Severity Index (PASI) Score at Week 52
Description: PASI: Combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section(head: 0.1, arms: 0.2 body: 0.3 legs: 0.4)
Time Frame: Week 40 , week 52
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned.
Measure: Number; unit: Percent of participants
Arm/Group | AIN457150 mg- Induction Period Only(IPO) | AIN457 300 mg - IPO | AIN457 150 mg - Fixed Interval (FI) | AIN457 300 mg FI | AIN457 150 mg- Start of Relapse (SoR) | AIN457 300 mg- SoR
Number analyzed (Participants) | 0 | 0 | 203 | 216 | 206 | 217
Percent of participants |  |  | 62.1 | 78.2 | 52.4 | 67.7

2. Secondary Outcome: Absolute Change From Baseline for PASI 50 / 75 / 90 / 100 and IGA 2011 Score of 0 or 1 at Week 2, 4, 6, 8, 12
Description: PASI: Combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section(head:01, arms:0.2 body:0.3 legs:0.4)
Time Frame: Baseline, week 2, 3 , 4, 8, 12
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AIN457150 mg- Induction Period Only(IPO) | AIN457 300 mg - IPO | AIN457 150 mg - Fixed Interval (FI) | AIN457 300 mg FI | AIN457 150 mg- Start of Relapse (SoR) | AIN457 300 mg- SoR
Number analyzed (Participants) | 482 | 483 | 0 | 0 | 0 | 0
Units on a scale
  Week 2 | -7.46 (6.338) | -9.28 (6.752) |  |  |  |
  Week 3 | -11.13 (7.826) | -12.97 (7.826) |  |  |  |
  Week 4 | -14.18 (8.956) | -15.90 (8.838) |  |  |  |
  Week 8 | -18.69 (10.147) | -19.56 (9.356) |  |  |  |
  Week 12 | -20.71 (10.804) | -20.89 (9.584) |  |  |  |

3. Secondary Outcome: Absolute Change From Baseline for PASI 50 / 75 / 90 / 100 and IGA 2011 Score of 0 or 1 at Week at Week 16, 20, 24,28,32,36,40,44,48,and Week 52
Description: as for outcome 2
Time Frame: Baseline, week 12,16,20,24,28,32,36,40,44,48 and week 52
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AIN457150 mg- Induction Period Only(IPO) | AIN457 300 mg - IPO | AIN457 150 mg - Fixed Interval (FI) | AIN457 300 mg FI | AIN457 150 mg- Start of Relapse (SoR) | AIN457 300 mg- SoR
Number analyzed (Participants) | 0 | 0 | 203 | 216 | 206 | 217
Units on a scale
  Week 12 |  |  | -21.52 (9.553) | -22.32 (8.943) | -23.19 (11.063) | -21.58 (9.448)
  Week 16 |  |  | -21.23 (9.676) | -22.61 (9.310) | -23.26 (11.158) | -21.58 (9.626)
  Week 20 |  |  | -20.79 (9.739) | -22.47 (9.237) | -22.28 (11.548) | -20.97 (9.787)
  Week 24 |  |  | -20.61 (9.745) | -22.30 (9.262) | -21.36 (11.938) | -20.09 (9.904)
  Week 28 |  |  | -20.29 (9.730) | -22.13 (9.244) | -20.53 (11.754) | -19.27 (9.844)
  Week 32 |  |  | -20.11 (9.847) | -21.98 (9.195) | -19.41 (10.962) | -18.68 (9.983)
  Week 36 |  |  | -19.82 (9.908) | -21.79 (9.324) | -18.86 (10.625) | -18.14 (9.352)
  Week 40 |  |  | -19.51 (9.821) | -21.71 (9.369) | -18.30 (10.660) | -17.89 (9.837)
  Week 44 |  |  | -19.40 (9.691) | -21.58 (9.398) | -17.73 (11.041) | -17.03 (9.876)
  Week 48 |  |  | -19.04 (10.093) | -21.34 (9.681) | -17.48 (10.638) | -16.58 (9.040)
  Week 52 |  |  | -18.79 (9.904) | 21.47 (9.402) | -17.40 (10.719) | -16.33 (8.322)

4. Secondary Outcome: Percent of Participants Achieving Psoriasis Area & Severity Index (PASI) Score and IGA Mod 2011 0 or 1 Score Over Time at Week 12 and 52 (Induction)
Description: PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4). PASI 50, 75, 90 and 100 were defined as participants achieving ≥ 50%, 75%, 90% or 100% improvement from baseline. The IGA mod 2011 scale is static, i.e. it referred exclusively to the participant's disease at the time of the assessment, and did not compare with any of the participant's previous disease states at previous visits. The scores are: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe
Time Frame: Baseline, week 2, 4, 6, 8, 12
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Number; unit: Percent of participant
Arm/Group | AIN457150 mg- Induction Period Only(IPO) | AIN457 300 mg - IPO | AIN457 150 mg - Fixed Interval (FI) | AIN457 300 mg FI | AIN457 150 mg- Start of Relapse (SoR) | AIN457 300 mg- SoR
Number analyzed (Participants) | 482 | 483 | 0 | 0 | 0 | 0
Percent of participant
  Week 2 IGA 0/1 | 1.2 | 3.1 |  |  |  |
  Week 2 PASI 75 | 1.9 | 5.2 |  |  |  |
  Week 2 PASI 50 | 20.2 | 32.9 |  |  |  |
  Week 2 PASI 90 | 0 | 0.2 |  |  |  |
  Week 2 PASI 100 | 0 | 0.2 |  |  |  |
  Week 3 IGA 0/1 | 5.2 | 9.3 |  |  |  |
  Week 3 PASI 75 | 11 | 19.3 |  |  |  |
  Week 3 PASI 50 | 43 | 63.6 |  |  |  |
  Week 3 PASI 90 | 1.5 | 3.1 |  |  |  |
  Week 3 PASI 100 | 0 | 0.6 |  |  |  |
  Week 4 IGA 0/1 | 15.6 | 25.5 |  |  |  |
  Week 4 PASI 75 | 27.9 | 42.9 |  |  |  |
  Week 4 PASI 50 | 66.3 | 81.8 |  |  |  |
  Week 4 PASI 90 | 6.7 | 13.7 |  |  |  |
  Week 4 PASI 100 | 0.4 | 2.3 |  |  |  |
  Week 8 IGA 0/1 | 47.8 | 59.4 |  |  |  |
  Week 8 PASI 75 | 63.8 | 76.8 |  |  |  |
  Week 8 PASI 50 | 88.4 | 93 |  |  |  |
  Week 8 PASI 90 | 32.4 | 45.8 |  |  |  |
  Week 8 PASI 100 | 8.3 | 13.9 |  |  |  |
  Week 12 IGA 0/1 | 62.8 | 76 |  |  |  |
  Week 12 PASI 75 | 84.4 | 90.1 |  |  |  |
  Week 12 PASI 50 | 93.1 | 96.1 |  |  |  |
  Week 12 PASI 90 | 49.3 | 64.2 |  |  |  |
  Week 12 PASI 100 | 16.2 | 25.7 |  |  |  |

5. Secondary Outcome: Percent of Participants Achieving Psoriasis Area & Severity Index (PASI) Score and IGA Mod 2011 0 or 1 Score Over Time at Week 12 and 52 (Maintenance Period))
Description: The IGA mod 2011 is a static scale, i.e., it refers exclusively to the participant's disease state at the time of the assessments and does not attempt a comparison to any of the participant's previous disease states at prior visits. The score ranges from 0 (clear) to 4 (severe. The score 0 is clear, 1 is almost clear, 2 is mild, 3 is moderate, and 4 is severe
Time Frame: Baseline, week 16,20,24,28,32,36,40,44,48, and Week 52
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Number; unit: Percent of participants
Arm/Group | AIN457150 mg- Induction Period Only(IPO) | AIN457 300 mg - IPO | AIN457 150 mg - Fixed Interval (FI) | AIN457 300 mg FI | AIN457 150 mg- Start of Relapse (SoR) | AIN457 300 mg- SoR
Number analyzed (Participants) | 0 | 0 | 203 | 216 | 206 | 217
Percent of participants
  Week 16 IGA 0/1 |  |  | 70.9 | 82.4 | 74.8 | 83.4
  Week 16 PASI 75 |  |  | 90.1 | 92.1 | 92.7 | 94.9
  Week 16 PASI 50 |  |  | 96.1 | 97.7 | 98.1 | 98.2
  Week 16 PASI 90 |  |  | 59.1 | 75.5 | 68.4 | 76.5
  Week 16 PASI 100 |  |  | 27.6 | 31.5 | 22.3 | 38.2
  Week 20 IGA 0/1 |  |  | 69 | 75.5 | 64.6 | 77
  Week 20 PASI 75 |  |  | 85.7 | 90.3 | 81.6 | 87.1
  Week 20 PASI 50 |  |  | 94.6 | 97.7 | 92.2 | 97.2
  Week 20 PASI 90 |  |  | 62.6 | 74.5 | 55.8 | 72.8
  Week 20 PASI 100 |  |  | 29.1 | 35.6 | 24.8 | 35.5
  Week 24 IGA 0/1 |  |  | 67.5 | 76.9 | 56.3 | 65.9
  Week 24 PASI 75 |  |  | 80.3 | 88 | 72.3 | 77.9
  Week 24 PASI 50 |  |  | 93.1 | 94.9 | 89.3 | 94
  Week 24 PASI 90 |  |  | 66.5 | 74.1 | 51.5 | 59.9
  Week 24 PASI 100 |  |  | 29.1 | 36.1 | 19.9 | 26.3
  Week 28 IGA 0/1 |  |  | 65.5 | 72.7 | 44.7 | 52.5
  Week 28 PASI 75 |  |  | 77.3 | 85.6 | 65 | 71.4
  Week 28 PASI 50 |  |  | 92.6 | 93.5 | 87.4 | 94
  Week 28 PASI 90 |  |  | 60.6 | 70.4 | 40.8 | 50.2
  Week 28 PASI 100 |  |  | 29.6 | 38 | 15.5 | 23
  Week 32 IGA 0/1 |  |  | 64 | 74.1 | 33.5 | 46.1
  Week 32 PASI 75 |  |  | 74.9 | 84.3 | 50.5 | 63.1
  Week 32 PASI 50 |  |  | 91.1 | 92.6 | 82 | 90.3
  Week 32 PASI 90 |  |  | 58.6 | 74.1 | 32.5 | 41.5
  Week 32 PASI 100 |  |  | 30.5 | 38.9 | 10.7 | 15.7
  Week 36 IGA 0/1 |  |  | 59.6 | 70.4 | 27.2 | 33.6
  Week 36 PASI 75 |  |  | 71.4 | 82.9 | 45.1 | 58.1
  Week 36 PASI 50 |  |  | 87.7 | 91.2 | 78.6 | 94
  Week 36 PASI 90 |  |  | 54.7 | 68.1 | 24.8 | 35.5
  Week 36 PASI 100 |  |  | 28.6 | 38.9 | 2.9 | 7.4
  Week 40 IGA 0/1 |  |  | 53.2 | 68.5 | 26.2 | 35.5
  Week 40 PASI 75 |  |  | 68 | 81.5 | 42.2 | 58.5
  Week 40 PASI 50 |  |  | 87.7 | 90.7 | 74.8 | 88.9
  Week 40 PASI 90 |  |  | 52.2 | 68.5 | 18.9 | 26.7
  Week 40 PASI 100 |  |  | 26.1 | 38 | 1.9 | 7.4
  Week 44 IGA 0/1 |  |  | 52.7 | 64.8 | 20.4 | 27.6
  Week 44 PASI 75 |  |  | 66 | 80.1 | 37.4 | 51.2
  Week 44 PASI 50 |  |  | 84.2 | 92.1 | 72.8 | 82.5
  Week 44 PASI 90 |  |  | 49.8 | 66.2 | 16.5 | 22.1
  Week 44 PASI 100 |  |  | 22.7 | 39.8 | 1.5 | 4.6
  Week 48 IGA 0/1 |  |  | 51.7 | 64.8 | 20.4 | 21.7
  Week 48 PASI 75 |  |  | 65.5 | 78.7 | 33 | 45.6
  Week 48 PASI 50 |  |  | 83.3 | 89.8 | 74.8 | 82
  Week 48 PASI 90 |  |  | 49.8 | 62.5 | 12.6 | 14.7
  Week 48 PASI 100 |  |  | 21.2 | 38.4 | 1 | 3.7
  Week 52 IGA 0/1 |  |  | 47.3 | 59.3 | 18 | 20.3
  Week 52 PASI 75 |  |  | 62.1 | 78.2 | 35 | 41
  Week 52 PASI 50 |  |  | 83.7 | 87.5 | 73.8 | 81.1
  Week 52 PASI 90 |  |  | 45.8 | 59.7 | 11.2 | 13.8
  Week 52 PASI 100 |  |  | 21.2 | 36.6 | 2.4 | 5.1

6. Secondary Outcome: Change From Baseline in EQ-5D at Each Visit, up to Week 52, (Induction)
Description: ED-5Q: Participant rated questionnaire to assess health related quality of life in terms of a single utility score. Five domains are assessed mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each with three possible score: 1 indicates no problems, better state of health; 3 indicates worst state of health (example "confined to bed") A visual analog scale (VAS) assesses the health status from 0 (worst possible health state) to 100 (best possible health state)
Time Frame: Baseline to week 2, 4, 8, 12
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AIN457150 mg- Induction Period Only(IPO) | AIN457 300 mg - IPO | AIN457 150 mg - Fixed Interval (FI) | AIN457 300 mg FI | AIN457 150 mg- Start of Relapse (SoR) | AIN457 300 mg- SoR
Number analyzed (Participants) | 482 | 483 | 0 | 0 | 0 | 0
Units on a scale
  Week 2 | 5.9 (14.64) | 7.6 (12.86) |  |  |  |
  Week 4 | 10.8 (17.79) | 13.6 (18.63) |  |  |  |
  Week 8 | 17.5 (20.79) | 18.3 (21.51) |  |  |  |
  Week 12 | 20.2 (23.47) | 21.2 (24.08) |  |  |  |

7. Secondary Outcome: Change From Baseline in EQ-5D at Each Visit, up to Week 52, (Maintenance)
Description: as for outcome 6
Time Frame: Baseline to week 16, 20, 24, 28, 32, 36, 40, 44, 48, and Week 52.
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AIN457150 mg- Induction Period Only(IPO) | AIN457 300 mg - IPO | AIN457 150 mg - Fixed Interval (FI) | AIN457 300 mg FI | AIN457 150 mg- Start of Relapse (SoR) | AIN457 300 mg- SoR
Number analyzed (Participants) | 0 | 0 | 203 | 216 | 206 | 217
Units on a scale
  Week 16 |  |  | 21.4 (25.11) | 23 (22.44) | 23.4 (25.31) | 23.9 (26.09)
  Week 20 |  |  | 20.6 (25.07) | 23 (23.27) | 22.1 (26.04) | 22.4 (27.45)
  Week 24 |  |  | 20.6 (25.05) | 22.9 (23.32) | 20 (26.66) | 22.3 (26.47)
  Week 28 |  |  | 19.4 (26.46) | 23 (22.71) | 19.3 (25.07) | 20.4 (26.26)
  Week 32 |  |  | 20.4 (24.95) | 22.8 (23.22) | 17.9 (24.97) | 18.8 (25.90)
  Week 36 |  |  | 19.6 (25.79) | 23 (22.67) | 17.4 (24.30) | 17.7 (26.15)
  Week 40 |  |  | 19.8 (25.39) | 22.8 (22.69) | 16.3 (23.53) | 16.4 (26.38)
  Week 44 |  |  | 19.8 (25.53) | 22.3 (23.10) | 15.4 (23.70) | 14.9 (26.81)
  Week 48 |  |  | 19.7 (25.33) | 22.7 (22.85) | 16.2 (23.17) | 13.4 (26.65)
  Week 52 |  |  | 18.3 (25.63) | 23 (22.40) | 16.7 (23.30) | 13.4 (25.68)

8. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Score. up to Week 52, (Induction)
Description: The DLQI is a quality of life measure used in the psoriatic The 10-item questionnaire has a score range of 0 (best) to 30 (worst) with higher scores indicating poor quality of life. The instrument contains six functional scales (i.e., symptoms and feeling, daily activities, leisure, work and school, personal relationships, treatment). Each item has 4 response categories, ranging from 0 (not at all) to 3 (very much). "Not relevant" is also a valid response and is scored as 0. The DLQI total score is a sum of the 10 questions
Time Frame: Baseline to week 2, 4, 8, 12
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AIN457150 mg- Induction Period Only(IPO) | AIN457 300 mg - IPO | AIN457 150 mg - Fixed Interval (FI) | AIN457 300 mg FI | AIN457 150 mg- Start of Relapse (SoR) | AIN457 300 mg- SoR
Number analyzed (Participants) | 482 | 483 | 0 | 0 | 0 | 0
Units on a scale
  Week 2 DLQI total score | -5.5 (5.02) | -6 (5.10) |  |  |  |
  Week 4 DLQI total score | -8.2 (6.11) | -8.7 (6.29) |  |  |  |
  Week 8 DLQI total score | -10.2 (6.40) | -10.3 (6.73) |  |  |  |
  Week 12 DLQI total score | -10.8 (6.75) | -11 (7.01) |  |  |  |

9. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Score. up to Week 52, (Maintenance)
Description: as for outcome 8
Time Frame: Baseline to week 16, 20, 24, 28, 32, 36, 40, 44, 48, and Week 52.
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AIN457150 mg- Induction Period Only(IPO) | AIN457 300 mg - IPO | AIN457 150 mg - Fixed Interval (FI) | AIN457 300 mg FI | AIN457 150 mg- Start of Relapse (SoR) | AIN457 300 mg- SoR
Number analyzed (Participants) | 0 | 0 | 203 | 216 | 206 | 217
Units on a scale
  Week 16 |  |  | -11 (6.63) | -11.4 (7.12) | -11.4 (6.98) | -11.3 (7.58)
  Week 20 |  |  | -10.6 (6.50) | -11 (7.18) | -10.6 (7.55) | -11 (7.64)
  Week 24 |  |  | -10.5 (6.67) | -11.1 (7.39) | -10.1 (7.65) | -10.3 (7.71)
  Week 28 |  |  | -10.5 (6.68) | -11 (7.22) | -9.7 (7.39) | -9.5 (7.46)
  Week 32 |  |  | -10.5 (6.76) | -10.9 (7.17) | -8.6 (7.66) | -8.9 (7.61)
  Week 36 |  |  | -10.2 (6.94) | -10.9 (7.30) | -8.6 (7.55) | -8.5 (7.79)
  Week 40 |  |  | -10.1 (6.83) | -10.8 (7.33) | -8.4 (7.22) | -8.5 (7.59)
  Week 44 |  |  | -10.2 (6.72) | -10.8 (7.46) | -8.4 (7.07) | -8.6 (7.29)
  Week 48 |  |  | -10 (6.57) | -10.8 (7.38) | -8.6 (7.41) | 7.9 (7.02)
  Week 52 |  |  | -9.8 (7.06) | -10.9 (7.31) | -8.4 (7.46) | -7.6 (7.14)

10. Secondary Outcome: % of Participants Achieving a DLQI Score of 0 or 1 at Each Visit up to Week 52, (Induction)
Description: as for outcome 8
Time Frame: Baseline to week 2, 4, 6, 8, 12
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Number; unit: Percent of participants
Arm/Group | AIN457150 mg- Induction Period Only(IPO) | AIN457 300 mg - IPO | AIN457 150 mg - Fixed Interval (FI) | AIN457 300 mg FI | AIN457 150 mg- Start of Relapse (SoR) | AIN457 300 mg- SoR
Number analyzed (Participants) | 482 | 484 | 0 | 0 | 0 | 0
Percent of participants
  Week 2 (n=463,471) | 9.5 | 13.8 |  |  |  |
  Week 4 (n=479,482) | 23.2 | 33.2 |  |  |  |
  Week 8 (n=479,482) | 44.7 | 52.1 |  |  |  |
  Week 12 (n=479,482) | 53.4 | 63.1 |  |  |  |

11. Secondary Outcome: % of Participants Achieving a DLQI Score of 0 or 1 at Each Visit up to Week 52, (Maintenance).
Description: as for outcome 8
Time Frame: Baseline to week 16, 20, 24, 28, 32, 36, 40, 44, 48, and Week 52
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Number; unit: Percent of participant
Arm/Group | AIN457150 mg- Induction Period Only(IPO) | AIN457 300 mg - IPO | AIN457 150 mg - Fixed Interval (FI) | AIN457 300 mg FI | AIN457 150 mg- Start of Relapse (SoR) | AIN457 300 mg- SoR
Number analyzed (Participants) | 0 | 0 | 203 | 216 | 206 | 217
Percent of participant
  Week 16 (n=199,209,202,215) |  |  | 59.8 | 66.5 | 58.4 | 72.1
  Week 20 (n=202,213,205,217) |  |  | 57.4 | 67.6 | 58 | 69.6
  Week 24 (n=202,214,206,217) |  |  | 58.4 | 68.7 | 53.9 | 65.4
  Week 28 (n=202,214,206,217) |  |  | 57.9 | 70.1 | 47.6 | 51.6
  Week 32 (n=202,214,206,217) |  |  | 57.9 | 67.8 | 37.9 | 47.5
  Week 36 (n=202,214,206,217) |  |  | 58.4 | 65 | 39.8 | 39.6
  Week 40 (n=202,214,206,217) |  |  | 55 | 66.4 | 35 | 42.4
  Week 44 (n=202,214,206,217) |  |  | 59.9 | 68.7 | 31.6 | 43.3
  Week 48 (n=202,214,206,217) |  |  | 54 | 67.3 | 32 | 40.6
  Week 52 (n=202,214,206,217) |  |  | 56.4 | 69.2 | 31.1 | 37.3

12. Secondary Outcome: Median Time to Relapse (Weeks) From Week 12.
Description: Median time to relapse (weeks) from week 12. Relapse is defined as greater than 50% loss of the maximal PASI improvement from baseline. PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4). A negative mean percentage change indicates improvement
Time Frame: Week 12 to week 16, 20, 24, 28, 32, 36, 40, 44, 48, and Week 52.
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Median (95% Confidence Interval); unit: Number of weeks
Arm/Group | AIN457150 mg- Induction Period Only(IPO) | AIN457 300 mg - IPO | AIN457 150 mg - Fixed Interval (FI) | AIN457 300 mg FI | AIN457 150 mg- Start of Relapse (SoR) | AIN457 300 mg- SoR
Number analyzed (Participants) | 0 | 0 | 203 | 216 | 206 | 217
Number of weeks |  |  | NA [NA to NA] — not estimable due to insufficient events at the time of analysis | NA [NA to NA] — not estimable due to insufficient events at the time of analysis | NA [NA to NA] — not estimable due to insufficient events at the time of analysis | 302 [302 to NA] — not estimable due to insufficient events at the time of analysis

13. Secondary Outcome: Percent of Responders With PASI Equal to or Greater Than 50, PASI 75, PASI 90, PASI 100 and Percent of Responders With IGA Score of 0 or 1 Who Failed to Respond to a Previous Biologic Psoriasis Therapy
Description: as for outcome 4
Time Frame: Week 12
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned, only participants with evaluable data were included
Measure: Number; unit: Percent of participants
Arm/Group | AIN457150 mg- Induction Period Only(IPO) | AIN457 300 mg - IPO | AIN457 150 mg - Fixed Interval (FI) | AIN457 300 mg FI | AIN457 150 mg- Start of Relapse (SoR) | AIN457 300 mg- SoR
Number analyzed (Participants) | 64 | 74 | 0 | 0 | 0 | 0
Percent of participants
  Week 12 IGA 0/1 | 42.2 | 62.2 |  |  |  |
  Week 12 PASI 50 | 87.5 | 90.5 |  |  |  |
  Week 12 PASI 75 | 68.8 | 86.5 |  |  |  |
  Week 12 PASI 90 | 26.6 | 56.8 |  |  |  |
  Week 12 PASI 100 | 6.3 | 21.6 |  |  |  |

14. Secondary Outcome: Percent of Responders With PASI Equal to or Greater Than 50, PASI 75, PASI 90, PASI 100 and Percent of Responders With IGA Score of 0 or 1 Who Failed to Respond to a Previous Biologic Psoriasis Therapy
Description: as for outcome 4
Time Frame: Week 52
Population: as for outcome 13
Measure: Number; unit: Percent of participants
Arm/Group | AIN457150 mg- Induction Period Only(IPO) | AIN457 300 mg - IPO | AIN457 150 mg - Fixed Interval (FI) | AIN457 300 mg FI | AIN457 150 mg- Start of Relapse (SoR) | AIN457 300 mg- SoR
Number analyzed (Participants) | 0 | 0 | 21 | 36 | 23 | 28
Percent of participants
  Week 52 IGA 0/1 |  |  | 42.9 | 66.7 | 4.3 | 14.3
  Week 52 PASI 50 |  |  | 81 | 86.1 | 60.9 | 75
  Week 52 PASI 75 |  |  | 47.6 | 77.8 | 21.7 | 32.1
  Week 52 PASI 90 |  |  | 33.3 | 66.7 | 13 | 7.1
  Week 52 PASI 100 |  |  | 28.6 | 52.8 | 0 | 3.6

15. Secondary Outcome: Number of Visits With PASI 50, 75, 90, 100 Score and IGA Mod 2011 0 or 1
Description: as for outcome 4
Time Frame: Week 16, 20, 24,28,32,36,40,44,48,and Week 52
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Number; unit: Percent of participants
Arm/Group | AIN457150 mg- Induction Period Only(IPO) | AIN457 300 mg - IPO | AIN457 150 mg - Fixed Interval (FI) | AIN457 300 mg FI | AIN457 150 mg- Start of Relapse (SoR) | AIN457 300 mg- SoR
Number analyzed (Participants) | 0 | 0 | 203 | 216 | 206 | 217
Percent of participants
  PASI 50 Visit 0 |  |  | 1.5 | 0.9 | 0.5 | 0.5
  PASI 50 Visit 1 |  |  | 1 | 0.5 | 1.5 | 0.5
  PASI 50 Visit 2 |  |  | 2.5 | 0.5 | 3.4 | 0.5
  PASI 50 Visit 3 |  |  | 0.5 | 1.9 | 3.4 | 0.5
  PASI 50 Visit 4 |  |  | 1.5 | 2.8 | 4.4 | 1.8
  PASI 50 Visit 5 |  |  | 3.4 | 0.5 | 2.4 | 1.8
  PASI 50 Visit 6 |  |  | 2.5 | 0.5 | 4.9 | 0.9
  PASI 50 Visit 7 |  |  | 3 | 3.2 | 6.8 | 5.5
  PASI 50 Visit 8 |  |  | 3 | 1.9 | 10.2 | 12.4
  PASI 50 Visit 9 |  |  | 8.4 | 7.9 | 8.7 | 16.6
  PASI 50 Visit 10 |  |  | 72.9 | 79.6 | 53.9 | 59
  PASI 75 Visit 0 |  |  | 4.9 | 3.2 | 3.9 | 2.8
  PASI 75 Visit 1 |  |  | 5.9 | 2.8 | 6.8 | 2.3
  PASI 75 Visit 2 |  |  | 5.4 | 2.8 | 8.3 | 4.1
  PASI 75 Visit 3 |  |  | 3 | 3.2 | 7.8 | 6.9
  PASI 75 Visit 4 |  |  | 4.9 | 1.9 | 11.2 | 8.3
  PASI 75 Visit 5 |  |  | 3.4 | 1.9 | 10.7 | 10.6
  PASI 75 Visit 6 |  |  | 4.9 | 1.9 | 11.7 | 8.3
  PASI 75 Visit 7 |  |  | 4.4 | 3.7 | 9.2 | 11.1
  PASI 75 Visit 8 |  |  | 2.5 | 4.2 | 9.7 | 18.4
  PASI 75 Visit 9 |  |  | 7.4 | 8.8 | 10.7 | 15.2
  PASI 75 Visit 10 |  |  | 53.2 | 65.7 | 10.2 | 12
  PASI 90 Visit 0 |  |  | 24.6 | 12 | 23.8 | 15.7
  PASI 90 Visit 1 |  |  | 4.4 | 5.1 | 15 | 7.8
  PASI 90 Visit 2 |  |  | 2.5 | 3.7 | 8.3 | 12
  PASI 90 Visit 3 |  |  | 5.4 | 4.2 | 6.8 | 11.1
  PASI 90 Visit 4 |  |  | 4.4 | 2.3 | 11.2 | 11.1
  PASI 90 Visit 5 |  |  | 3.9 | 1.4 | 8.7 | 6.5
  PASI 90 Visit 6 |  |  | 3.4 | 5.1 | 9.7 | 8.8
  PASI 90 Visit 7 |  |  | 3.9 | 4.6 | 7.3 | 10.6
  PASI 90 Visit 8 |  |  | 5.4 | 6.5 | 2.9 | 8.3
  PASI 90 Visit 9 |  |  | 13.8 | 13.4 | 2.9 | 3.7
  PASI 90 Visit 10 |  |  | 28.1 | 41.7 | 3.4 | 4.6
  PASI 100 Visit 0 |  |  | 53.2 | 41.2 | 65 | 51.2
  PASI 100 Visit 1 |  |  | 5.9 | 6.5 | 9.7 | 7.8
  PASI 100 Visit 2 |  |  | 5.9 | 4.2 | 6.3 | 12.4
  PASI 100 Visit 3 |  |  | 3.4 | 4.6 | 7.3 | 8.8
  PASI 100 Visit 4 |  |  | 3.4 | 2.3 | 6.3 | 6.9
  PASI 100 Visit 5 |  |  | 3 | 5.6 | 2.9 | 6.5
  PASI 100 Visit 6 |  |  | 4.9 | 5.1 | 1 | 1.8
  PASI 100 Visit 7 |  |  | 4.4 | 3.7 | 0.5 | 2.3
  PASI 100 Visit 8 |  |  | 2.5 | 5.6 | 0 | 0.9
  PASI 100 Visit 9 |  |  | 4.4 | 7.9 | 0 | 0.5
  PASI 100 Visit 10 |  |  | 8.9 | 13.4 | 1 | 0.9
  IGA mod 2011 0 or 1 response Visit 0 |  |  | 19.2 | 11.6 | 20.4 | 12
  IGA mod 2011 0 or 1 response Visit 1 |  |  | 5.4 | 3.7 | 10.2 | 6.5
  IGA mod 2011 0 or 1 response Visit 2 |  |  | 2 | 3.7 | 9.7 | 7.4
  IGA mod 2011 0 or 1 response Visit 3 |  |  | 5.4 | 5.1 | 9.2 | 10.6
  IGA mod 2011 0 or 1 response Visit 4 |  |  | 3.9 | 3.2 | 8.3 | 12
  IGA mod 2011 0 or 1 response Visit 5 |  |  | 3.4 | 1.9 | 10.2 | 13.8
  IGA mod 2011 0 or 1 response Visit 6 |  |  | 6.4 | 4.6 | 9.2 | 7.8
  IGA mod 2011 0 or 1 response Visit 7 |  |  | 6.4 | 3.7 | 7.8 | 10.1
  IGA mod 2011 0 or 1 response Visit 8 |  |  | 5.9 | 2.8 | 5.8 | 8.3
  IGA mod 2011 0 or 1 response Visit 9 |  |  | 6.4 | 12.5 | 3.9 | 6
  IGA mod 2011 0 or 1 response Visit 10 |  |  | 35.5 | 47.2 | 5.3 | 5.5

16. Secondary Outcome: Number of Secukinumab Injections Needed to Regain PASI 75 Response From Start of Relapse After Week 12
Description: The number of secukinumab injections needed for participants to regain PASI 75 response from the start of relapse after week 12
Time Frame: week 16, 20, 24,28,32,36,40,44,48,and Week 52
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Number; unit: percent of participants
Arm/Group | AIN457150 mg- Induction Period Only(IPO) | AIN457 300 mg - IPO | AIN457 150 mg - Fixed Interval (FI) | AIN457 300 mg FI | AIN457 150 mg- Start of Relapse (SoR) | AIN457 300 mg- SoR
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 176 | 185
percent of participants
  SoR: one, Regain PASI 75 Injection 0 (n=97,128) |  |  |  |  | 4.1 | 0.8
  SoR: one, Regain PASI 75 Injection 1 (n=97,128) |  |  |  |  | 40.2 | 0
  SoR: one, Regain PASI 75 Injection 2 (n=97,128) |  |  |  |  | 27.8 | 45.3
  SoR: one, Regain PASI 75 Injection 3 (n=97,128) |  |  |  |  | 11.3 | 0
  SoR: one, Regain PASI 75 Injection 4 (n=97,128) |  |  |  |  | 6.2 | 31.3
  SoR: one, Regain PASI 75 Injection 5 (n=97,128) |  |  |  |  | 4.1 | 0
  SoR: one, Regain PASI 75 Injection 6 (n=97,128) |  |  |  |  | 4.1 | 14.1
  SoR: one, Regain PASI 75 Injection 7 (n=97,128) |  |  |  |  | 1 | 0
  SoR: one, Regain PASI 75 Injection 8 (n=97,128) |  |  |  |  | 1 | 3.1
  SoR: one, Regain PASI 75 Injection 10 (n=97,128) |  |  |  |  | 0 | 3.9
  SoR: one, Regain PASI 75 Injection 12 (n=97,128) |  |  |  |  | 0 | 1.6
  SoR: Two, Regain PASI 75 Injection 0 (n=21,36) |  |  |  |  | 0 | 5.6
  SoR: Two, Regain PASI 75 Injection 1 (n=21,36) |  |  |  |  | 47.6 | 0
  SoR: Two, Regain PASI 75 Injection 2 (n=21,36) |  |  |  |  | 42.9 | 58.3
  SoR: Two, Regain PASI 75 Injection 3 (n=21,36) |  |  |  |  | 4.8 | 0
  SoR: Two, Regain PASI 75 Injection 4 (n=21,36) |  |  |  |  | 0 | 19.4
  SoR: Two, Regain PASI 75 Injection 6 (n=21,36) |  |  |  |  | 4.8 | 8.3
  SoR: Two, Regain PASI 75 Injection 8 (n=21,36) |  |  |  |  | 0 | 8.3
  SoR: Three, Regain PASI 75 Injection 2 (n=0,4) |  |  |  |  | NA — No evaluable participants | 100

17. Secondary Outcome: Number of Participants Developing Anti-secukinumab Antibodies
Description: The development of anti-secunimubab anti-bodies will decrease a participant's ability to respond to secukinumab treatment. The number of participants developing anti-secukinumab anti-bodies was measured from Baseline to week 12, 24, 52 and 8 weeks after treatment at week 60
Time Frame: Baseline, weeks 12, 24, 52 and 60
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Number; unit: Number of participants
Arm/Group | AIN457150 mg- Induction Period Only(IPO) | AIN457 300 mg - IPO | AIN457 150 mg - Fixed Interval (FI) | AIN457 300 mg FI | AIN457 150 mg- Start of Relapse (SoR) | AIN457 300 mg- SoR
Number analyzed (Participants) | 0 | 0 | 203 | 216 | 206 | 217
Number of participants |  |  | 2 | 1 | 1 | 1

ADVERSE EVENTS:
Groups:
- INDUCTION-AIN457 150mg: INDUCTION-AIN457 150mg
- INDUCTION-AIN457 300mg: INDUCTION-AIN457 300mg
- ENTIRE-AIN457 150mg: ENTIRE-AIN457 150mg
- ENTIRE-AIN457 300mg: ENTIRE-AIN457 300mg
- ENTIRE-AIN457 150 mg SoR: ENTIRE-AIN457 150 mg SoR
- ENTIRE-AIN457 300 mg SoR: ENTIRE-AIN457 300 mg SoR
- FOLLOW UP-AIN457 150mg IPO: FOLLOW UP-AIN457 150mg IPO
- FOLLOW UP-AIN457 300mg IPO: FOLLOW UP-AIN457 300mg IPO
- FOLLOW UP-AIN457 150 mg: FOLLOW UP-AIN457 150 mg
- FOLLOW UP-AIN457 300 mg: FOLLOW UP-AIN457 300 mg
- FOLLOW UP-AIN457 150 mg SoR: FOLLOW UP-AIN457 150 mg SoR
- FOLLOW UP-AIN457 300 mg SoR: FOLLOW UP-AIN457 300 mg SoR
Arm/Group | INDUCTION-AIN457 150mg | INDUCTION-AIN457 300mg | ENTIRE-AIN457 150mg | ENTIRE-AIN457 300mg | ENTIRE-AIN457 150 mg SoR | ENTIRE-AIN457 300 mg SoR | FOLLOW UP-AIN457 150mg IPO | FOLLOW UP-AIN457 300mg IPO | FOLLOW UP-AIN457 150 mg | FOLLOW UP-AIN457 300 mg | FOLLOW UP-AIN457 150 mg SoR | FOLLOW UP-AIN457 300 mg SoR
Serious Adverse Events (participants affected / at risk) | 8/482 | 10/484 | 12/203 | 18/217 | 12/205 | 14/217 | 1/27 | 0/23 | 2/40 | 1/39 | 1/39 | 0/35
Other Adverse Events (participants affected / at risk) | 190/482 | 178/484 | 134/203 | 137/217 | 120/205 | 126/217 | 6/27 | 6/23 | 8/40 | 7/39 | 13/39 | 9/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | INDUCTION-AIN457 150mg (N=482) | INDUCTION-AIN457 300mg (N=484) | ENTIRE-AIN457 150mg (N=203) | ENTIRE-AIN457 300mg (N=217) | ENTIRE-AIN457 150 mg SoR (N=205) | ENTIRE-AIN457 300 mg SoR (N=217) | FOLLOW UP-AIN457 150mg IPO (N=27) | FOLLOW UP-AIN457 300mg IPO (N=23) | FOLLOW UP-AIN457 150 mg (N=40) | FOLLOW UP-AIN457 300 mg (N=39) | FOLLOW UP-AIN457 150 mg SoR (N=39) | FOLLOW UP-AIN457 300 mg SoR (N=35)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ANGINA PECTORIS (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
AORTIC VALVE INCOMPETENCE (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CORONARY ARTERY STENOSIS (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
PALPITATIONS (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FIBROUS DYSPLASIA OF BONE (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYDROCELE (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
VESTIBULAR DISORDER (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CROHN'S DISEASE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ILEUS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PANCREATITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GENERALISED OEDEMA (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HEPATIC STEATOSIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
HEPATITIS (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HEPATOTOXICITY (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LIVER INJURY (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
PORTAL HYPERTENSION (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
ABSCESS BACTERIAL (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ABSCESS OF SALIVARY GLAND (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
APPENDICITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
CELLULITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
CHRONIC TONSILLITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
GROIN ABSCESS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HELICOBACTER GASTRITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HEPATITIS B (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
INFLUENZA (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OOPHORITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PHARYNGEAL ABSCESS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PNEUMONIA VIRAL (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
POST PROCEDURAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SEPSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
TONSILLITIS BACTERIAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
VULVAL ABSCESS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CONCUSSION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
PANCREATIC INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
POST-TRAUMATIC PAIN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
SPINAL CORD INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
URINE ANALYSIS ABNORMAL (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GOUT (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
CHONDROMALACIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FRACTURE NONUNION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BENIGN BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
PITUITARY TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CENTRAL NERVOUS SYSTEM INFLAMMATION (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HAEMORRHAGIC STROKE (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPOAESTHESIA (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MULTIPLE SCLEROSIS (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SCIATICA (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
SYNCOPE (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
VASCULAR HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ALCOHOL ABUSE (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
ALCOHOL WITHDRAWAL SYNDROME (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ALCOHOLISM (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DEPRESSION (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PANIC ATTACK (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CALCULUS URETERIC (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
IGA NEPHROPATHY (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RENAL COLIC (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RENAL TUBULAR NECROSIS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
METRORRHAGIA (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
VARICOCELE (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
VULVA CYST (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DERMAL CYST (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PEMPHIGUS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PUSTULAR PSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GRANULOMATOSIS WITH POLYANGIITIS (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PERIPHERAL ARTERY STENOSIS (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | INDUCTION-AIN457 150mg (N=482) | INDUCTION-AIN457 300mg (N=484) | ENTIRE-AIN457 150mg (N=203) | ENTIRE-AIN457 300mg (N=217) | ENTIRE-AIN457 150 mg SoR (N=205) | ENTIRE-AIN457 300 mg SoR (N=217) | FOLLOW UP-AIN457 150mg IPO (N=27) | FOLLOW UP-AIN457 300mg IPO (N=23) | FOLLOW UP-AIN457 150 mg (N=40) | FOLLOW UP-AIN457 300 mg (N=39) | FOLLOW UP-AIN457 150 mg SoR (N=39) | FOLLOW UP-AIN457 300 mg SoR (N=35)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
CATARACT (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
CONJUNCTIVITIS (Eye disorders) | 0 | 3 | 3 | 5 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
ABDOMINAL TENDERNESS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 2 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 2 | 0 | 3 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 7 | 8 | 6 | 7 | 8 | 10 | 0 | 0 | 0 | 0 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 | 4 | 5 | 4 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
HYPERCHLORHYDRIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 10 | 4 | 5 | 3 | 5 | 1 | 0 | 0 | 0 | 0 | 1 | 0
TOOTHACHE (Gastrointestinal disorders) | 3 | 0 | 4 | 1 | 4 | 2 | 0 | 1 | 0 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 2 | 3 | 2 | 5 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
ASTHENIA (General disorders) | 1 | 3 | 1 | 0 | 2 | 3 | 0 | 0 | 1 | 0 | 0 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
INJECTION SITE PAIN (General disorders) | 3 | 4 | 0 | 4 | 3 | 5 | 0 | 0 | 0 | 0 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 4 | 4 | 4 | 3 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 0
PYREXIA (General disorders) | 3 | 0 | 4 | 5 | 5 | 2 | 0 | 0 | 2 | 0 | 3 | 0
BRONCHITIS (Infections and infestations) | 3 | 6 | 11 | 7 | 1 | 7 | 1 | 0 | 0 | 0 | 0 | 0
EAR INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
FOLLICULITIS (Infections and infestations) | 3 | 3 | 2 | 6 | 3 | 6 | 1 | 0 | 0 | 0 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 5 | 2 | 7 | 5 | 4 | 5 | 0 | 0 | 0 | 0 | 0 | 0
HERPES ZOSTER (Infections and infestations) | 3 | 1 | 3 | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0
INFLUENZA (Infections and infestations) | 6 | 6 | 9 | 6 | 5 | 8 | 1 | 0 | 0 | 0 | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 48 | 46 | 37 | 36 | 32 | 42 | 0 | 1 | 1 | 0 | 0 | 1
ORAL HERPES (Infections and infestations) | 3 | 2 | 2 | 2 | 4 | 2 | 0 | 0 | 0 | 1 | 0 | 0
PERIODONTITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 1
PHARYNGITIS (Infections and infestations) | 4 | 9 | 8 | 12 | 2 | 7 | 0 | 0 | 0 | 0 | 0 | 0
PHARYNGITIS BACTERIAL (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0
RHINITIS (Infections and infestations) | 5 | 3 | 4 | 6 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0
SINUSITIS (Infections and infestations) | 5 | 3 | 3 | 6 | 7 | 4 | 0 | 0 | 0 | 1 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 17 | 17 | 16 | 16 | 11 | 14 | 0 | 0 | 0 | 2 | 0 | 0
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 3 | 3 | 4 | 0 | 5 | 0 | 0 | 1 | 0 | 0 | 0
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 4 | 3 | 4 | 1 | 5 | 3 | 0 | 0 | 0 | 0 | 0 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 5 | 0 | 3 | 1 | 4 | 0 | 0 | 2 | 0 | 0 | 0 | 0
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 5 | 2 | 2 | 1 | 6 | 1 | 0 | 0 | 0 | 0 | 0 | 0
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 5 | 5 | 3 | 5 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 2 | 2 | 2 | 6 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 9 | 9 | 8 | 11 | 12 | 13 | 0 | 0 | 0 | 0 | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 10 | 4 | 12 | 9 | 9 | 7 | 0 | 0 | 0 | 0 | 0 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 1 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 6 | 2 | 5 | 4 | 6 | 2 | 0 | 0 | 1 | 0 | 0 | 0
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 4 | 1 | 5 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
SEBORRHOEIC KERATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 22 | 17 | 14 | 11 | 14 | 11 | 1 | 0 | 0 | 0 | 0 | 1
PARAESTHESIA (Nervous system disorders) | 1 | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
INSOMNIA (Psychiatric disorders) | 9 | 1 | 6 | 1 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0
DYSURIA (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
GLYCOSURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
KETONURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 10 | 10 | 13 | 11 | 8 | 8 | 0 | 0 | 1 | 0 | 1 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 3 | 10 | 3 | 7 | 0 | 0 | 0 | 0 | 0 | 0
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 5 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 5 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 2 | 1 | 3 | 5 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 1 | 6 | 0 | 8 | 1 | 7 | 0 | 0 | 0 | 0 | 0 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0
ERYTHRODERMIC PSORIASIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 3 | 4 | 5
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 20 | 12 | 12 | 13 | 17 | 6 | 0 | 0 | 0 | 1 | 2 | 1
PSORIASIS (Skin and subcutaneous tissue disorders) | 1 | 7 | 0 | 3 | 1 | 6 | 0 | 0 | 0 | 1 | 1 | 0
PUSTULAR PSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 2
SEBORRHOEIC DERMATITIS (Skin and subcutaneous tissue disorders) | 4 | 2 | 5 | 6 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 3 | 4 | 6 | 2 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 11 | 11 | 9 | 17 | 9 | 12 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
A limitation of this study is the lack of a placebo group; however, because the placebo response is very low in psoriasis, it is inappropriate to maintain patients on placebo for 52 weeks. .

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety